CLINICAL TRIAL: NCT07194616
Title: Impact of Neoadjuvant Chemoradiotherapy Versus Surgery Alone on Circulating Tumor Cells in Patients With Stage II-III Rectal Cancer and Negative Circumferential Resection Margin: a Multicenter Randomized Clinical Trial
Brief Title: Rectal Cancer CTC Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Palacky University (Other); University Hospital Olomouc (Other); Municipal Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECTA-CTC
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer Patients
Keywords: circulating tumor cells; liquid biopsy; neoadjuvant chemoradiotherapy; prognostic biomarkers; rectal cancer; surgical resection
MeSH Terms: conditions — Neoplastic Cells, Circulating; Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Surgery (Experimental): Procedure: rectal resection with TME (Total Mesorectal Excision)
  Interventions: Procedure: Primary Surgery
- Neoadjuvant radiochemotherapy and surgery (Experimental): Procedure: rectal resection with TME performed 6-10 weeks after completion of chemoradiotherapy.
  Interventions: Procedure: Neoadjuvant radiochemotherapy and surgery

INTERVENTIONS:
Procedure: Primary Surgery — Patients undergo radical surgical resection with TME without preceding neoadjuvant therapy
  Arms: Primary Surgery
Procedure: Neoadjuvant radiochemotherapy and surgery — Neoadjuvant treatment: long-course pelvic radiotherapy (conventional fractionation) with concurrent chemotherapy (standard fluoropyrimidine-based regimen)
  Arms: Neoadjuvant radiochemotherapy and surgery

SUMMARY:
This prospective, multi-centre, randomised clinical trial aims to compare the effect of neoadjuvant chemoradiotherapy versus primary surgery on circulating tumor cells (CTCs) in patients with stage II-III rectal cancer without circumferential resection mar-gin involvement. CTCs are considered a promising biomarker for disease dissemination and treatment response. Patients will be randomized to either primary surgical resection with total mesorectal excision or long-course neoadjuvant chemoradiotherapy followed by surgery. Serial blood samples will be collected at predefined time points to assess the presence and dynamics of CTCs. Secondary endpoints include perioperative morbidity and mortality, local recurrence rate, disease-free survival, and overall survival. The results of this study may provide new insights into the prognostic role of CTCs and contribute to optimising treatment strategies for rectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer remains one of the most common malignancies worldwide, and rectal cancer requires a multidisciplinary treatment approach. For patients with locally advanced rectal cancer, neoadjuvant chemoradiotherapy (nCRT) followed by surgical resection has been widely used to reduce the risk of local recurrence. However, the indication for nCRT in patients without circumferential resection margin (CRM) involvement remains controversial. While some studies have suggested benefits of nCRT, others have shown comparable oncological outcomes with primary surgery when high-quality total mesorectal excision (TME) is performed.

Circulating tumor cells (CTCs) are malignant cells detectable in peripheral blood that have been associated with metastatic potential and poor prognosis in various cancers, including colorectal cancer. Monitoring the presence and dynamics of CTCs offers a minimally invasive "liquid biopsy" approach that may provide prognostic information and reflect treatment efficacy. Existing evidence suggests that changes in CTC levels after surgery or systemic therapy may correlate with recurrence risk and survival, but relevant data in rectal cancer patients undergoing multimodal treatment are limited.

This prospective, multi-centre, randomised clinical trial will enrol patients with stage II-III rectal cancer without evidence of CRM involvement on staging magnetic resonance imaging (MRI). Eligible patients will be randomized into two study arms:

1. Primary surgery arm: radical surgical resection with total mesorectal excision (TME).
2. Neoadjuvant therapy arm: long-course neoadjuvant chemoradiotherapy fol-lowed by delayed surgical resection.

Peripheral blood samples will be collected at predefined time points in both groups to determine the presence and quantity of CTCs. The primary objective is to compare the effect of neoadjuvant chemoradiotherapy versus surgery alone on CTC dynamics.

Secondary objectives include:

* Evaluation of short-term surgical outcomes (perioperative complications, 30-day morbidity and mortality).
* Assessment of long-term oncological outcomes (local recurrence, disease-free survival, and overall survival at 3 and 5 years).

By integrating CTC monitoring into a modern randomized clinical trial design, this study aims to clarify the prognostic value of CTCs in rectal cancer and determine whether specific treatment strategies are associated with more favourable biological and clinical outcomes. The findings may contribute to more individualised treatment planning and potentially reduce the risk of recurrence and mortality in rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed rectal adenocarcinoma within 12 cm from anal verge
* Stage II (cT3-4 N0 M0) or stage III (cT1-4 N1-2, M0)
* Negative circumferential resection margin on staging MRI
* ASA physical status I-III
* Signed informed consent

Exclusion Criteria:

* Tumor infiltration beyond fascia recti propria on MRI
* Metastatic disease (stage IV)
* Recurrent rectal cancer
* Other concurrent malignancies
* Emergency surgery required
* Contraindication to surgery under general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Circulating Tumor Cells (CTC) Dynamics - neoadjuvant treatment - shape | (1) before the initiation of CRT, (2) 1 week and (3) 1 month after the initiation of CRT, (4) preoperatively (1-2 weeks before surgery), (5) 1 week postoperatively, and (6) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of CTC round shape will be observed.
Circulating Tumor Cells (CTC) Dynamics - neoadjuvant treatment - size | (1) before the initiation of CRT, (2) 1 week and (3) 1 month after the initiation of CRT, (4) preoperatively (1-2 weeks before surgery), (5) 1 week postoperatively, and (6) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The CTC size will be observed, with the border value of > 4 μm.
Circulating Tumor Cells (CTC) Dynamics - neoadjuvant treatment - DAPI positivity | (1) before the initiation of CRT, (2) 1 week and (3) 1 month after the initiation of CRT, (4) preoperatively (1-2 weeks before surgery), (5) 1 week postoperatively, and (6) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The DAPI positivity will be observed. A DAPI-positive nucleus is a cell nucleus that has been stained with DAPI (4',6-diamidino-2-phenylindole), a fluorescent dye that binds specifically to the adenine-thymine (A-T) rich regions of double-stranded DNA.
Circulating Tumor Cells (CTC) Dynamics - neoadjuvant treatment - pancytokeratin and/or EpCAM positivity | (1) before the initiation of CRT, (2) 1 week and (3) 1 month after the initiation of CRT, (4) preoperatively (1-2 weeks before surgery), (5) 1 week postoperatively, and (6) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of pancytokeratin and/or EpCAM positivity in CTCs will be observed. EpCAM positivity refers to the presence of EpCAM (Epithelial Cell Adhesion Molecule) protein on cells, which is a marker primarily expressed on epithelial cells and in many carcinomas.
Circulating Tumor Cells (CTC) Dynamics - neoadjuvant treatment - CD45 negativity | (1) before the initiation of CRT, (2) 1 week and (3) 1 month after the initiation of CRT, (4) preoperatively (1-2 weeks before surgery), (5) 1 week postoperatively, and (6) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of CD45 negativity in CTCs will be observed. "CD45 negative" means a cell does not express the CD45 protein on its surface.
Circulating Tumor Cells (CTC) Dynamics - primary surgery - shape | (1) preoperatively (1-2 weeks before surgery), (2) 1 week postoperatively, and (3) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of CTC round shape will be observed.
Circulating Tumor Cells (CTC) Dynamics - primary surgery - size | (1) preoperatively (1-2 weeks before surgery), (2) 1 week postoperatively, and (3) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The CTC size will be observed, with the border value of > 4 μm.
Circulating Tumor Cells (CTC) Dynamics - primary surgery - DAPI positivity | (1) preoperatively (1-2 weeks before surgery), (2) 1 week postoperatively, and (3) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The DAPI positivity will be observed. A DAPI-positive nucleus is a cell nucleus that has been stained with DAPI (4',6-diamidino-2-phenylindole), a fluorescent dye that binds specifically to the adenine-thymine (A-T) rich regions of double-stranded DNA.
Circulating Tumor Cells (CTC) Dynamics - primary surgery - pancytokeratin and/or EpCAM positivity | (1) preoperatively (1-2 weeks before surgery), (2) 1 week postoperatively, and (3) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of pancytokeratin and/or EpCAM positivity in CTCs will be observed. EpCAM positivity refers to the presence of EpCAM (Epithelial Cell Adhesion Molecule) protein on cells, which is a marker primarily expressed on epithelial cells and in many carcinomas.
Circulating Tumor Cells (CTC) Dynamics - primary surgery - CD45 negativity | (1) preoperatively (1-2 weeks before surgery), (2) 1 week postoperatively, and (3) 1 month postoperatively
  The detection of CTC in laboratory will be performed using fluorescence microscope. Potential CTC candidates (hotspots) were identified based on green fluorescence and subjected to operator review. The presence of CD45 negativity in CTCs will be observed. "CD45 negative" means a cell does not express the CD45 protein on its surface.

SECONDARY OUTCOMES:
Short-term postoperative outcomes - preoperative complications | Within 30 days after surgery
  The occurrence of perioperative complications will be observed
Short-term postoperative outcomes - 30-day morbidity | Within 30 days after surgery
  30-day morbidity will be observed
Short-term postoperative outcomes - 30-day mortality | Within 30 days after surgery
  30-day mortality will be observed
Local recurrence rate | Up to 5 years
  Cumulative incidence of local tumor recurrence after treatment.
Disease-free survival (DFS) | 3 and 5 years after surgery
  Interval from treatment to recurrence, progression, or death.
Overall survival (OS) | 3 and 5 years after surgery
  Proportion of patients alive at 3 and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ihnát, prof., MD, PhD, MBA, Principal Investigator — University Hospital Ostrava
Locations (4):
- Czechia (4):
  - University Hospital Olomouc, Olomouc
  - Palacky University Olomouc, Faculty of Medicine, Olomouc
  - University Hospital Ostrava, Ostrava
  - Municipal Hospital Ostrava - Fifejdy, Ostrava

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon reasonable request.

REFERENCES:
- [Background] Lu CY, Uen YH, Tsai HL, Chuang SC, Hou MF, Wu DC, Juo SH, Lin SR, Wang JY. Molecular detection of persistent postoperative circulating tumour cells in stages II and III colon cancer patients via multiple blood sampling: prognostic significance of detection for early relapse. Br J Cancer. 2011 Mar 29;104(7):1178-84. doi: 10.1038/bjc.2011.40. Epub 2011 Feb 22. PMID 21343933
- [Background] Hinz S, Roder C, Tepel J, Hendricks A, Schafmayer C, Becker T, Kalthoff H. Cytokeratin 20 positive circulating tumor cells are a marker for response after neoadjuvant chemoradiation but not for prognosis in patients with rectal cancer. BMC Cancer. 2015 Dec 16;15:953. doi: 10.1186/s12885-015-1989-z. PMID 26674974
- [Background] Yadav A, Kumar A, Siddiqui MH. Detection of circulating tumour cells in colorectal cancer: Emerging techniques and clinical implications. World J Clin Oncol. 2021 Dec 24;12(12):1169-1181. doi: 10.5306/wjco.v12.i12.1169. PMID 35070736
- [Background] Burz C, Pop VV, Buiga R, Daniel S, Samasca G, Aldea C, Lupan I. Circulating tumor cells in clinical research and monitoring patients with colorectal cancer. Oncotarget. 2018 May 11;9(36):24561-24571. doi: 10.18632/oncotarget.25337. eCollection 2018 May 11. PMID 29849961
- [Background] Wu J, Li Z, Zou J, Li L, Cui N, Hao T, Yi K, Yang J, Wu Y. A meta-analysis of the value of circulating tumor cells in monitoring postoperative recurrence and metastasis of colorectal cancer. PLoS One. 2022 Sep 19;17(9):e0274282. doi: 10.1371/journal.pone.0274282. eCollection 2022. PMID 36121855
- [Background] Sun W, Li G, Wan J, Zhu J, Shen W, Zhang Z. Circulating tumor cells: A promising marker of predicting tumor response in rectal cancer patients receiving neoadjuvant chemo-radiation therapy. Oncotarget. 2016 Oct 25;7(43):69507-69517. doi: 10.18632/oncotarget.10875. PMID 27486758
- [Background] Pan RJ, Hong HJ, Sun J, Yu CR, Liu HS, Li PY, Zheng MH. Detection and Clinical Value of Circulating Tumor Cells as an Assisted Prognostic Marker in Colorectal Cancer Patients. Cancer Manag Res. 2021 Jun 8;13:4567-4578. doi: 10.2147/CMAR.S300554. eCollection 2021. PMID 34135633
- [Background] Tseng M, Soon YY, Vellayappan B, Ho F, Tey J. Radiation therapy for rectal cancer. J Gastrointest Oncol. 2019 Dec;10(6):1238-1250. doi: 10.21037/jgo.2018.12.04. PMID 31949945
- [Background] Uen YH, Lu CY, Tsai HL, Yu FJ, Huang MY, Cheng TL, Lin SR, Wang JY. Persistent presence of postoperative circulating tumor cells is a poor prognostic factor for patients with stage I-III colorectal cancer after curative resection. Ann Surg Oncol. 2008 Aug;15(8):2120-8. doi: 10.1245/s10434-008-9961-7. Epub 2008 May 15. PMID 18481151
- [Background] Kulu Y, Tarantino I, Billeter AT, Diener MK, Schmidt T, Buchler MW, Ulrich A. Comparative Outcomes of Neoadjuvant Treatment Prior to Total Mesorectal Excision and Total Mesorectal Excision Alone in Selected Stage II/III Low and Mid Rectal Cancer. Ann Surg Oncol. 2016 Jan;23(1):106-13. doi: 10.1245/s10434-015-4832-5. Epub 2015 Aug 25. PMID 26305025
- [Background] Rahbari NN, Elbers H, Askoxylakis V, Motschall E, Bork U, Buchler MW, Weitz J, Koch M. Neoadjuvant radiotherapy for rectal cancer: meta-analysis of randomized controlled trials. Ann Surg Oncol. 2013 Dec;20(13):4169-82. doi: 10.1245/s10434-013-3198-9. Epub 2013 Sep 4. PMID 24002536
- [Background] Ihnat P, Zidlik V, Ihnat Rudinska L, Koscielnik P, Hanzlikova P, Skarda J. Magnetic resonance imaging in preoperative assessment of the mesorectal nodal status of patients with rectal cancer - Can it be trusted? Eur J Radiol. 2023 Aug;165:110961. doi: 10.1016/j.ejrad.2023.110961. Epub 2023 Jul 5. PMID 37423017
- [Background] Sauer R, Fietkau R, Wittekind C, Rodel C, Martus P, Hohenberger W, Tschmelitsch J, Sabitzer H, Karstens JH, Becker H, Hess C, Raab R; German Rectal Cancer Group. Adjuvant vs. neoadjuvant radiochemotherapy for locally advanced rectal cancer: the German trial CAO/ARO/AIO-94. Colorectal Dis. 2003 Sep;5(5):406-15. doi: 10.1046/j.1463-1318.2003.00509.x. PMID 12925071
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv263. doi: 10.1093/annonc/mdy161. No abstract available. PMID 29741565
- [Background] van de Velde CJ, Boelens PG, Tanis PJ, Espin E, Mroczkowski P, Naredi P, Pahlman L, Ortiz H, Rutten HJ, Breugom AJ, Smith JJ, Wibe A, Wiggers T, Valentini V. Experts reviews of the multidisciplinary consensus conference colon and rectal cancer 2012: science, opinions and experiences from the experts of surgery. Eur J Surg Oncol. 2014 Apr;40(4):454-68. doi: 10.1016/j.ejso.2013.10.013. Epub 2013 Nov 8. PMID 24268926
- [Background] Ihnat P, Srovnal J, Stejskal P, Vidlarova M, Skacelikova E, Snajder B, Varga A, Ihnat Rudinska L. Monitoring Treatment Response in Rectal Cancer through Circulating Tumor Cell Dynamics: A Pilot Clinical Study. J Surg Oncol. 2025 Nov;132(6):1052-1057. doi: 10.1002/jso.70073. Epub 2025 Sep 2. PMID 40891187